CLINICAL TRIAL: NCT04344275
Title: The Immediate Effects of Kinesio-Taping on Scapular Muscle Endurance and Strength in Asymptomatic Subjects: A Single-Blind, Randomized, Placebo-Controlled Study
Brief Title: The Immediate Effects of Kinesio-Taping on Scapular Muscle Endurance and Strength in Asymptomatic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Zeynep Hazar Kanik, Associate professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 25901600-537
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Asymptomatic Subjects
Keywords: Kinesio-taping; Scapula; Endurance; Muscle strength; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio-taping (KT) (Experimental): The skin will first be properly cleaned with rubbing alcohol. An I-shaped strip of Kinesio tape with a 5-cm width was applied over the middle trapezius from origin to insertion in the KT group. Kinesio-tape size was measured from the T3 spinal process to the acromion, while the subject is in sitting position relaxed with the arm at the trunk side. The subject was then instructed to move the arm into horizontal adduction and neck flexion. At this position, the tape was applied involving the middle trapezius, ending on the acromion, with 50% tension as recommended for this technique.
  Interventions: Other: -Scapular endurance test; Other: -Muscle strength test
- Placebo Kinesio-taping (KT) (Placebo Comparator): Kinesio-tape was applied with no tension and technique on the middle trapezius.
  Interventions: Other: -Scapular endurance test; Other: -Muscle strength test

INTERVENTIONS:
Other: -Scapular endurance test — The resistance of the trapezius and serratus anterior muscles to fatigue was assessed using the scapular muscle endurance test.
Other: -Muscle strength test — Upper trapezius (UT), middle trapezius (MT), lower trapezius (LT), and serratus anterior (SA) muscle strengths were tested using a hand-held digital dynamometer (Lafayette Manual Muscle Tester, Model 01165).

SUMMARY:
The purpose of this study was to investigate the immediate effects of Kinesio-taping (KT) on scapular muscle endurance and strength and compared to placebo Kinesio-taping in asymptomatic subjects.

DETAILED DESCRIPTION:
Thirty-nine asymptomatic subjects (20 females and 19 males, mean age 20.46±1.09 years, mean BMI 21.99±3.02 kg/m2) were included in this study. Subjects were randomly allocated to KT (with the muscle facilitation technique) and placebo-KT (without any technique and tension). Scapular isometric muscle endurance was measured with a scapular muscle endurance test. The strength of the upper, middle, and lower trapezius, and serratus anterior was assessed using a hand-held digital dynamometer. Data were analyzed with 2x2 [groups (KT and Placebo-KT) x time (pre- and post-intervention)] mixed-model ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* An age range of 18 to 25 years,
* The ability to participate voluntarily.

Exclusion Criteria:

* Shoulder injuries in the last year, previous shoulder surgery, shoulder dislocation, and having performed upper-body exercises within the 24 hours before each evaluation session. - Diagnosed with cardiovascular or neurological disease

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Scapular endurance test | 1 day
  The resistance of the trapezius and serratus anterior muscles to fatigue was assessed using the scapular muscle endurance test. Subjects were in standing position with their shoulders and elbows flexed to 90°, and they were instructed to hold a dynamometer between their hands. The scapula was placed in a neutral position, and an adjustable spacer was set between their elbows to maintain the test position. Then, the subjects were asked to externally rotate the shoulders to attain a 1-kg load and to maintain this force, which was displayed on the dynamometer. The test was terminated when the subjects were unable to maintain the resistance and dropped the adjustable spacer, failed to maintain the 90° shoulder flexion, or reported an unbearable discomfort. The test was carried out twice and the average result recorded in seconds.
Muscle strength test | 1 day
  Upper trapezius (UT), middle trapezius (MT), lower trapezius (LT), and serratus anterior (SA) muscle strengths were tested using a hand-held digital dynamometer (Lafayette Manual Muscle Tester, Model 01165). Strength of these muscles was assessed with the "break test method," in which the subject resisted the prescribed motion until the examiner overcame the subject's isometric contraction. Test position of trapezius and serratus anterior muscles was described by Ekstrom et al. Following a familiarization test, subjects performed two trials with standardized verbal encouragement, and the average value of the 2 trials was used for statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep HAZAR KANIK, PhD, PT, Study Chair — Gazi University
Locations (1):
- Gazi University, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No